CLINICAL TRIAL: NCT04163822
Title: Clinical Characteristics and Outcome Analysis of Bronchopulmonary Dysplasia in Premature Infants With Typical Imaging Changes
Brief Title: Analysis of BPD in Premature Infants With Typical Imaging Changes
Status: Completed | Type: Observational
Sponsor: Wang Jianhui (Other)
Responsible Party: Sponsor-Investigator, Wang Jianhui, Attending doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 00020190209
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; typical chest imaging findings; clinical characteristics; outcomes; preterm infants; propensity score
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group with typical imaging changes: the BPD infants with typical chest imaging findings include fibrotic opacities and cysts on CXR or CT scans during the entire hospital stay.
  Interventions: Other: no intervention
- group without typical imaging changes: the infants meet the diagnosis criteria of BPD, but lack of typical chest imaging findings
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, only observation

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a common chronic respiratory disease in preterm infants. The increase in the survival rate of premature babies following the improvement of perinatal treatment and care has caused an increase in the incidence of BPD in recent years, which has seriously affected the quality of life of preterm infants. According to the consensus reached at the workshop sponsored by the National Institute of Child Health and Human Development (NICHD) in 2001, BPD was clinically defined based on oxygen dependency in preterm infants. However, the refined NICHD definition of BPD in 2018 emphasizes imaging findings to support a diagnosis of lung parenchyma disease.

Fibrotic opacities and cystic changes on chest imaging (chest X-ray [CXR] or computed tomography [CT] scan) were considered typical findings in BPD patients. In patients with severe BPD, the presence of bubbles/cystic appearance on CXR after 28 days of life was reported to be an important factor, and typical imaging findings can predict a poor pulmonary outcome in BPD patients. BPD is associated with poor outcomes. Although many studies have been conducted on BPD, there are limited reports specifically evaluating the association of typical imaging findings with clinical characteristics and later outcomes in patients with BPD.

We hypothesized that BPD with typical imaging findings was likely to be a particular subgroup of this entity, with a unique etiology, clinical characteristics and prognosis. Therefore, this retrospective study aimed to compare clinical characteristics, short-term outcomes and follow-up data until 2 years of age in preterm infants with or without typical imaging findings of BPD on CXR or CT scan during the entire hospital stay. A propensity score analysis was used to reduce bias between the two groups, and multivariate logistic regression analysis was performed to identify factors related to mortality in preterm infants with BPD.

ELIGIBILITY:
inclusion criteria: (1) BPD diagnosis according to the 2001 NICHD consensus; (2) chest imaging examination (CXR or CT) in the first week after birth; and (3) hospitalization within the first 7 days after birth.

exclusion criteria: (1) major congenital malformations or laboratory-confirmed chromosomal abnormalities; (2) inadequate clinical data or missing chest imaging data; or (3) loss to follow-up.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 9036 preterm infants with GA <36 weeks were admitted to the Department of Neonatology, CHCMU, from January 1, 2014, to December 31, 2018. Among them, 399 (4.4%) infants were diagnosed with BPD. Then, infants who were hospitalized after 7 days of life with missing data and lost to follow-up were excluded. Ultimately, 256 preterm infants were enrolled; 78 (30.5%) had typical chest imaging findings, whereas 178 (69.5%) did not have typical imaging findings. After PSM, the matched groups consisted of 58 pairs of patients.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, M.D, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Department of Neonatology,Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Arai H, Ito T, Ito M, Ota S, Takahashi T; Neonatal Research Network of Japan. Impact of chest radiography-based definition of bronchopulmonary dysplasia. Pediatr Int. 2019 Mar;61(3):258-263. doi: 10.1111/ped.13786. Epub 2019 Mar 7. PMID 30636380
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Kim HR, Kim JY, Yun B, Lee B, Choi CW, Kim BI. Interstitial pneumonia pattern on day 7 chest radiograph predicts bronchopulmonary dysplasia in preterm infants. BMC Pediatr. 2017 May 15;17(1):125. doi: 10.1186/s12887-017-0881-1. PMID 28506211
- [Background] Kim DH, Choi CW, Kim EK, Kim HS, Kim BI, Choi JH, Lee MJ, Yang EG. Association of increased pulmonary interleukin-6 with the priming effect of intra-amniotic lipopolysaccharide on hyperoxic lung injury in a rat model of bronchopulmonary dysplasia. Neonatology. 2010 Jun;98(1):23-32. doi: 10.1159/000263056. Epub 2009 Dec 2. PMID 19955834
- [Background] Choi CW, Lee J, Oh JY, Lee SH, Lee HJ, Kim BI. Protective effect of chorioamnionitis on the development of bronchopulmonary dysplasia triggered by postnatal systemic inflammation in neonatal rats. Pediatr Res. 2016 Feb;79(2):287-94. doi: 10.1038/pr.2015.224. Epub 2015 Nov 9. PMID 26551413
- [Background] Viscardi RM, Hasday JD. Role of Ureaplasma species in neonatal chronic lung disease: epidemiologic and experimental evidence. Pediatr Res. 2009 May;65(5 Pt 2):84R-90R. doi: 10.1203/PDR.0b013e31819dc2f9. PMID 19190528
- [Background] Lowe J, Watkins WJ, Edwards MO, Spiller OB, Jacqz-Aigrain E, Kotecha SJ, Kotecha S. Association between pulmonary ureaplasma colonization and bronchopulmonary dysplasia in preterm infants: updated systematic review and meta-analysis. Pediatr Infect Dis J. 2014 Jul;33(7):697-702. doi: 10.1097/INF.0000000000000239. PMID 24445836
- [Background] Steinhorn R, Davis JM, Gopel W, Jobe A, Abman S, Laughon M, Bancalari E, Aschner J, Ballard R, Greenough A, Storari L, Thomson M, Ariagno RL, Fabbri L, Turner MA; International Neonatal Consortium. Chronic Pulmonary Insufficiency of Prematurity: Developing Optimal Endpoints for Drug Development. J Pediatr. 2017 Dec;191:15-21.e1. doi: 10.1016/j.jpeds.2017.08.006. No abstract available. PMID 29173299
- [Derived] Ruan Q, Wang J, Shi Y. Clinical Characteristics and Outcomes Until 2 Years of Age in Preterm Infants With Typical Chest Imaging Findings of Bronchopulmonary Dysplasia: A Propensity Score Analysis. Front Pediatr. 2021 Aug 23;9:712516. doi: 10.3389/fped.2021.712516. eCollection 2021. PMID 34497783

RESULTS

PARTICIPANT FLOW:
Groups:
- Typical Imaging Findings (+): BPD infants with typical chest imaging findings( including fibrotic opacities and cysts on CXR or CT scans during the entire hospital stay.)
- Typical Imaging Findings (-): BPD infants without typical chest imaging findings
Period: Overall Study
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Started | 78 | 178
Completed | 78 | 178
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age means Gestational age(months)
Groups:
- Typical Imaging Finding (+): Infants with typical imaging findings
- Typical Imaging Finding (-): Infants without typical imaging findings
- Total: Total of all reporting groups
Arm/Group | Typical Imaging Finding (+) | Typical Imaging Finding (-) | Total
Number analyzed (Participants) | 78 | 178 | 256
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 29.4 [28 to 31.1] | 30.6 [29.4 to 31.1] | 30.3 [28.9 to 32.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 70 | 108
  Male | 40 | 108 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 78 | 178 | 256
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: the number of death/total number（%）
Time Frame: between 28 days after birth and 2 years of age
Population: number of each group after PSM
Measure: Count of Participants; unit: Participants
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 58 | 58
Participants | 17 | 7

2. Primary Outcome: Number of Participants According to the Severity of BPD
Description: Mild BPD: Breathing room air Moderate BPD: Need* for < 30% oxygen Severe BPD: Need* for ≥ 30% oxygen and/or positive pressure
Time Frame: 36 wk PMA(infants with GA>32w) or>28 d but <56 d(infants with GA>32w) or discharge to home, whichever comes first
Population: After psm,each group has 58 infants
Measure: Count of Participants; unit: Participants
Groups:
- Typical Imaging Findings (-): infants whitnout typical imaging findings
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 58 | 58
Participants
  severe BPD | 19 | 7
  mild-moderate BPD | 39 | 51

3. Primary Outcome: Number of Participants Who Need HOT at Discharge
Description: need of home oxygen therapy (HOT) at discharge
Time Frame: at discharge, an average of 2 months
Population: each group has 58 infants after PSM
Measure: Count of Participants; unit: Participants
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 58 | 58
Participants | 43 | 27

4. Secondary Outcome: Duration of Hospital Stay
Description: days between admission and first discharge
Time Frame: at discharge, an average of 2 months
Population: each group has 58 infants after PSM
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 58 | 58
days | 59 [33.8 to 68.2] | 56.5 [45.2 to 65.0]

5. Secondary Outcome: Routine Physical Assessment
Description: the measure of infant's length and weight: Underweight/Stunting Stunting was defined as >2 standard deviations (SD) below the mean length for age, and underweight was defined as >2 SD below the mean weight for age. Weight and length were calculated with Chinese growth reference standards
Time Frame: 2 Years of Age
Population: each group has 58 infants after PSM; 17 and 7 infants died in each group before they reached 2 years old.
Measure: Count of Participants; unit: Participants
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 41 | 51
Participants
  Underweight | 3 | 4
  Stunting | 4 | 7
  children without underweight and stunting | 34 | 40

6. Secondary Outcome: Days of Oxygen Supplement
Description: days during which the infants were given oxygen supplement
Time Frame: at discharge, an average of 46-56 days
Population: each group has 58 infants after PSM
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 58 | 58
days | 56 [32.7 to 68.2] | 46 [38 to 56.2]

7. Secondary Outcome: Wheezing Disorders
Description: Wheezing disorders were defined as a physician diagnosis of wheezing exposure treated with anti-asthma drugs (bronchodilators and corticosteroids)
Time Frame: between discharge and follow-up, an average of 22 months
Population: each group has 58 infants after PSM; 17 and 7 infants died in each group during the follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 41 | 51
Participants | 5 | 3

8. Secondary Outcome: Clinical Visits and Rehospitalizations
Description: clinical visits and rehospitalizations for a respiratory reason
Time Frame: between discharge and follow-up until 2 years of age, an average of 22 months
Population: each group has 58 infants after PSM; 17 infants and 7 infants died in each group during follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
Number analyzed (Participants) | 41 | 51
Participants
  Clinical visits <5 times | 20 | 33
  Clinical visits 5-10 times | 11 | 10
  Clinical visits >10 times | 10 | 8

ADVERSE EVENTS:
Time Frame: Admission date, 2 years
Arm/Group | Typical Imaging Findings (+) | Typical Imaging Findings (-)
All-Cause Mortality (participants affected / at risk) | 17/58 | 7/58
Serious Adverse Events (participants affected / at risk) | 19/58 | 7/58
Other Adverse Events (participants affected / at risk) | 4/78 | 6/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Typical Imaging Findings (+) (N=58) | Typical Imaging Findings (-) (N=58)
severe bpd (General disorders) | 19 (19) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Typical Imaging Findings (+) (N=78) | Typical Imaging Findings (-) (N=178)
leucomalacia (General disorders) | 4 (4) | 6 (6)

LIMITATIONS AND CAVEATS:
(1) this is a retrospective study, which inevitably leads to loss of follow-up and clinical data. A standardized follow-up program has not been perfected in our unit, especially 3 years ago or even earlier. (2) This is a single-center study of Chinese premature infants.(3) We used propensity score matching to balance some of the known confounding variables between the groups. However, it is inevitable to pay the cost of missing samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04163822/Prot_SAP_000.pdf